CLINICAL TRIAL: NCT03623802
Title: Integral Movement Therapy Versus Local Movement Therapy Approach in Patients With Idiopathic Chronic Low Back Pain: a Randomized Controlled Trail.
Brief Title: Integral Versus Local Movement Therapy Approach in Patients With Idiopathic Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Assoc. Prof. Dr. Sc., University of Primorska
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBPStudy-0120-93/2018/6
Record Dates: First submitted 2018-07-31; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Movement therapy; Supervised training
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The study design is a randomized clinical trial with parallel-group design including two intervention groups: integral movement therapy and conventional local movement therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Movement Therapy (Experimental): Group receiving treatment in form of Local Movement Therapy Program.
  Interventions: Other: Local Movement Therapy
- Integral Movement Therapy (Experimental): Group receiving treatment in form of Integral Movement Therapy Program.
  Interventions: Other: Integral Movement Therapy

INTERVENTIONS:
Other: Local Movement Therapy — Loads and intensity of exercises will be increased according to participants' abilities. Modifications of exercises are made through different body positions or increasing the load. When a participant will be able to perform a certain number of repetitions and sets of a required exercise, without any compensatory movements, he/she can proceed to the next level of exercise. Breaks between exercises and sets are the same as in the integral movement therapy protocol. Protocol consists of four basic exercises, which are progressed through sessions: (I) Abdomen curl. (II) Trunk extension on roman chair. (III) Hip bridge. (IV) Side plank.
  Arms: Local Movement Therapy
Other: Integral Movement Therapy — Protocol consists of four basic exercises, which are progressed through sessions: (I) Proprioception - sitting on an unstable surface - Swiss ball, with additional tasks with legs and arms. (II) Strength - pushing task in different body positions: a) Unstable position - from single plane to multi-plane arm movements. b) Stable position - high number of repetitions - single plane movement. (III) Strength - pulling task in different body positions: a) Unstable position - from single plane to multi-plane arm movements. b) Stable position - high number of repetitions - single plane movement. (IV) Lifting and carrying the loads: a) Stoop lifting. b) Squat lifting. c) Half kneeling lifting.
  Arms: Integral Movement Therapy

SUMMARY:
Systematic reviews evaluating the effectiveness of supervised exercise therapies commonly conclude that, to date, there is no evidence to support the superiority of one form of exercise over another. Randomized controlled trials to date included mostly trunk strengthening exercises (e.g. bird dog, plank) and there is no evidence about supervised, individually graded integral movement therapy program for patients with chronic low back pain (CLBP).

The research design is a randomized clinical trial with parallel-group design including two intervention groups: integral movement therapy and conventional local movement therapy. Participants in each group will receive 20 supervised sessions in a 10 week period, two times per week, with approximately 1 hour per session. Outcome assessments will occur at baseline and immediately post-intervention, follow up will take place at 6 months and 12 months after finishing the intervention. Pre specified analyses will evaluate the main effects of the treatment.

This trial will use a novel, previously unexplored integral approach to CLBP through exercises. In contrast to commonly used exercise programs, the integral program does not include specific local strength exercises for hip and trunk flexors and extensors. However, learning dynamic trunk muscle control in various body positions with added limb movements could be beneficial because of the parallels to everyday work. The study will contribute to clinical practice by providing evidence to guide professionals when deciding for the proper and efficient treatment of patients with CLBP.

DETAILED DESCRIPTION:
Literature suggests several different methods for coping with CLBP. Supervised exercise therapies are among the most commonly advocated treatments for nonspecific CLBP. However, findings from a systematic reviews concluded the most effective model of exercise therapy remain uncertain. Although several supervised randomized controlled trails, focusing on different approaches for managing the CLBP using movement therapy have been published so far, there is no evidence about integral movement therapy program for patients with CLBP. Systematic reviews evaluating the effectiveness of supervised exercise therapies commonly conclude that, to date, there is no evidence to support the superiority of one form of exercise over another. Randomized controlled trials to date include mostly trunk strengthening exercises (e.g. bird dog, plank).

The Primary study aim is to evaluate the efficiency of supervised and individually graded integral movement therapy program in patients with CLBP on pain, quality of life and functional abilities. Further, the secondary aim is to compare the difference in outcome measures to supervised, conventional local movement therapy. The following research questions are addressed:

(I) Does the supervised and individually graded integral movement therapy program have an effect on reducing pain, improving the quality of life and functional abilities in patients with chronic idiopathic low back pain? (II) Does the supervised and individually graded integral movement therapy program have a clinically more significant effect on reducing pain, improving the quality of life and functional abilities compared to the supervised, conventional local movement therapy? (III) Which program has a better effect on specific core stability strength (e.g., maximal isometric trunk flexion, extension and lateral flexion) and proprioception?

We intend to allocate 80 adults, aged between 30 and 60 years old, into two groups. Repeated measurements will be performed at the baseline and post therapy. Follow-up measures will take place 6 months and one year after the last therapy and include an International Physical Activity Questionnaire (IPAQ), qualitative and quantitative assessment of pain with the Oswestry disability index questionnaire (ODI) and the Numerical rating scale (NRS)

Eligibility Inclusion criteria

1. Chronic idiopathic low back pain which persists at least 12 weeks or two acute low back pain episodes in the last 12 months.
2. Patients aged between 30 and 60 years.
3. Capable of at least low physical activity to be able to complete movement therapy program.

Exclusion criteria

1. Severe spinal stenosis, spondylolisthesis, fibromyalgia.
2. Lumbar spine surgery.
3. Vascular disease.
4. Neurological deficits because of nerve root or spinal cord compression.
5. Ongoing treatment for low back pain.
6. Pregnancy.
7. Comorbid health conditions that could prevent active participation in exercise.

Participants in each group will receive 20 supervised sessions in 10 weeks' time, two times per week, with approximately 1 hour per session. Sessions will be carried out in small groups, up to 5 participants and will be supervised by an experienced kinesiologist or physiotherapist.

Both therapy programs start with general warm up on the elliptic trainer machine for 5 minutes, followed by specific warm up for the next 5 minutes including hip flexors, hip extensors and back extensors stretching. Each stretch is repeated once and held for 30 seconds. Part of the warm up routine is also learning the squat technique, pelvic neutral position and posture corrections. The Cool down routine includes same stretches as the warm up, with each stretch repeated twice (Additional file 3, part 1).

Each week, participants will receive a verbal quote of the week - back school. Quotes will be focused on posture, core activation and back position during lifting and carrying the loads, self-management of back pain, standing up and sitting down on the floor, pushing and pulling the objects and putting shoes on and off.

Each participant will be asked to keep his/her own exercise diary in order to follow the exercise intensity - body position, color of elastic, number of sets and repetitions in each set. Participant can move to the next level of exercise, when the required number of repetitions and sets are performed without any compensatory movements of the body and with complete core stability.

Integral movement therapy:

Load and intensity of exercises will be increased according to participants' abilities. Modifications of exercises are made by different body positions with decreasing the stability of body position or increasing elastic resistance. When a participant is able to perform a certain number of repetitions and sets of the required exercise, without any compensatory movements, he/she can proceed to the next level of exercise. There will be 1-2 minutes breaks between each exercise and 20 seconds breaks between sets of the same exercise. In the set break, participants will perform easy trunk motions (e.g.: hip circling, lateral flexion), to increase hydration of the intervertebral discs.

Protocol consists of four basic exercises, which are progressed through sessions (Additional file 3, part 2):

(I) Proprioception - sitting on an unstable surface - Swiss ball, with additional tasks with legs and arms.

(II) Strength - pushing task in different body positions:

1. Unstable position - from single plane to multi-plane arm movements.
2. Stable position - high number of repetitions - single plane movement. (III) Strength - pulling task in different body positions:

a) Unstable position - from single plane to multi-plane arm movements. b) Stable position - high number of repetitions - single plane movement. (IV) Lifting and carrying the loads:

1. Stoop lifting.
2. Squat lifting.
3. Half kneeling lifting.

Local movement therapy

Loads and intensity of exercises will be increased according to participants' abilities. Modifications of exercises are made through different body positions or increasing the load. When a participant is able to perform a certain number of repetitions and sets of a required exercise, without any compensatory movements, he/she can proceed to the next level of exercise. Breaks between exercises and sets are the same as in the integral movement therapy protocol.

Protocol consists of four basic exercises, which are progressed through sessions (Additional file 3, part 3):

(I) Abdomen curl. (II) Trunk extension on roman chair. (III) Hip bridge. (IV) Side plank.

There are two aspects of primary outcome measures. First part of the measures is based on different questionnaires: level of disability (ODI questionnaire), physical activity (IPAQ questionnaire) and pain (NRS questionnaire). All questionnaires will be conducted at baseline, immediately post-intervention, 6 months and 12 months after finishing the intervention, as medium and long-term follow-ups. Second part consists of different functional tests: timed up and go test (TUG), sit to stand test, chair seat and reach test (CSR), 6 minute walk test (6MW), Biering Sorensen test (BS), modified Schober test (mSCH) and Sharpened Romberg balance test (SRB). Those will be collected at baseline and immediately post-intervention.

The ODI questionnaire is one of the instruments for measuring disability caused by low back pain. The Slovenian version of the ODI questionnaire is a reliable and valid instrument for assessing outcomes of physical therapy in patients with chronic non-specific low back pain. IPAQ was developed as an instrument for cross-national monitoring of physical activity and inactivity and has reasonable measurement properties for monitoring population levels of physical activity among 18-65 years old adults in diverse settings. Pain intensity is frequently measured on an 11-point pain intensity numerical rating scale, where 0 means no pain and 10 is worst possible pain. On average, a reduction of two points or a reduction of approximately 30% in the NRS considered as a clinically important difference.

TUG test, sit to stand test, CSR and 6MW test are part of Senior Fitness Test battery. Specifically, the tests measure the level of physical abilities (strength, endurance, agility) that are impaired in patients with chronic low back pain.

Weak trunk muscles and reduced flexibility/elasticity of the back and hamstrings were found as a residual sign, in particular among those with recurrence or persistence of LBP. BS test provides reliable measures of position-holding time and can discriminate between subjects with and without nonspecific low back pain. Furthermore, literature states that mSCH test showed moderate validity and excellent reliability and metrically detected changes in sample of patients with CLBP. SRB has been reported to have good interrater reliability and test-retest reliability. Balance will be measured in three different positions of feet, parallel, semi tandem and tandem position, all with closed and opened eyes.

As this intervention requires no expensive equipment (elastic bands and Swiss ball, optional weights), it is suitable to perform at any physiotherapy or kinesiology department. What is more, when patients learn to perform the exercises, they can continue performing it at home with no extra costs. The study will contribute to clinical practice by providing evidence to guide professionals when deciding for the proper and efficient treatment of patients with CLBP. The results of this study will be published once the study is concluded

ELIGIBILITY:
Inclusion Criteria:

* Chronic idiopathic low back pain which persists at least 12 weeks or two acute low back pain episodes in the last 12 months.
* Patients aged between 30 and 60 years.
* Capable of at least low physical activity to be able to complete movement therapy program.

Exclusion Criteria:

* Severe spinal stenosis, spondylolisthesis, fibromyalgia.
* Lumbar spine surgery.
* Vascular disease.
* Neurological deficits because of nerve root or spinal cord compression.
* Ongoing treatment for low back pain.
* Pregnancy.
* Comorbid health conditions that could prevent active participation in exercise.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
CHANGE IN INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE (IPAQ) SCORE | 1 week before the first therapy, after 11 weeks, at 6-month follow up and at 12-month follow up.
  The International Physical Activity Questionnaire (IPAQ) is developed to measure health-related physical activity (PA) in populations.
Change in Oswestry Low Back Disability Questionnaire (ODI) Score | 1 week before the first therapy, after 11 weeks, at 6-month follow up and at 12-month follow up.
  Oswestry Low Back Disability Questionnaire is used to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.
Change inn Numeric Rating Scale for Pain (NRS) Score | 1 week before the first therapy, after 11 weeks, at 6-month follow up and at 12-month follow up.
  The NRS for pain is a unidimensional measure of pain intensity in adults.

SECONDARY OUTCOMES:
Change in Timed-up-and-go test (TUG) score | 1 week before the first therapy and after 11 weeks of therapy.
  TUG test measures physical function and correlates with fall risk.
Change in Sit-to-stand test score | 1 week before the first therapy and after 11 weeks of therapy.
  Sit-to-stand test is used to measure of lower limb strength and related function.
Change in Chair sit-and-reach test score | 1 week before the first therapy and after 11 weeks of therapy.
  The Chair Sit and Reach test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness. It is a variation of the traditional sit and reach flexibility test.
Change in 6 minute walk test score | 1 week before the first therapy and after 11 weeks of therapy.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in Spine flexibility. | 1 week before the first therapy and after 11 weeks of therapy.
  We will use the Schober's test, which is a physical examination used in physical medicine. to measure the ability of a patient to flex the lower back.
Change in Spinal extensor endurance | 1 week before the first therapy and after 11 weeks of therapy.
  The Biering-Sorensen test is used for evaluating the isometric endurance of the hip and back extensor muscles. Participant being tested gets on the therapeutic table in a horizontal prone position with their arms crossed over the chest, chin tucked, and the upper edge of the iliac crest on the pad. Once they are in this full position, the timer is started.
Change in Sharpened Romberg test score | 1 week before the first therapy and after 11 weeks of therapy.
  Sharpened Modified Romberg Test is used to assess postural stability. Participants stand in heel to toe position, with their arms folded across chest and eyes closed. The duration that they are able to maintain their balance is recorded. The test ceases at 30 sec or loss of balance (excessive sway, loss of balance, stepping during test, opening eyes).
Change in Trunk Muscle Strength | 1 week before the first therapy and after 11 weeks of therapy.
  Trunk Strength will be assessed by measuring maximal force that trunk muscles are able to exert in isometric conditions, on a custom-made dynamometer. Trunk extensors, flexors and lateroflexors will be tested.
Change in trunk reposition error test score | 1 week before the first therapy and after 11 weeks of therapy.
  In this test, participants are instructed to assume the position they are previously lead to. The difference between the position is described as the reposition error.
Change in maximal pelvic inclination | 1 week before the first therapy and after 11 weeks of therapy.
  Maximal pelvic inclination at full trunk flexion is an additional measure of lumbo-pelvic mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Šarabon, PhD, Principal Investigator — Faculty of Health Sciences, University of Primorska, Slovenia
Locations (1):
- Health Center Kranj, Kranj, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pustivsek S, Sarabon N. Integral movement therapy versus local movement therapy approach in patients with idiopathic chronic low-back pain: study protocol for a randomized controlled trial. Trials. 2019 Jan 21;20(1):69. doi: 10.1186/s13063-018-3128-z. PMID 30665438